CLINICAL TRIAL: NCT03508557
Title: Implementing Advance Care Planning Conversation Tools in Family Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Frailty Network (Other)
Responsible Party: Principal Investigator, Michelle Howard, Assistant Professor, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TG2015-03D
Record Dates: First submitted 2018-04-16; First posted 2018-04-25 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Frail Elderly Syndrome; Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: Single group before-after
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advance care planning tools (Experimental): Advance care planning education and structured conversation using tools
  Interventions: Behavioral: Advance care planning tools

INTERVENTIONS:
Behavioral: Advance care planning tools — Structured conversations between patients/substitute decision-maker and clinician based on education about advance care planning using locally relevant booklet/website, values clarification tool for patient engagement, clinician use of the Serious Illness Conversation Guide

SUMMARY:
This study evaluates the use of advance care planning conversation tools with patients attending their family doctor's office. Patients complete tools about their values and wishes, and a health care provider uses a structured discussion tool to talk about the patient's health condition and future wishes. The patient's family member/substitute decision-maker is encouraged to attend and be part of the discussions.

DETAILED DESCRIPTION:
Structured tools are helpful for advance care planning. Tools have been developed to help with advance care planning because it is a process which has multiple steps and people involved. This study will help health care teams in primary care learn to use the tools with frail or older seriously ill patients and will evaluate the perceptions of patients, family members and health care providers, as well as the impact of having the discussions on subsequent health care interactions the patient has.

Patients complete tools about their values and wishes, and a health care provider uses a structured discussion tool to talk about the patient's health condition and future wishes. The patient's family member/substitute decision-maker is encouraged to attend and be part of the discussions.

ELIGIBILITY:
Inclusion Criteria:

* age 60 or older
* chronic condition that may reduce life expectancy as per physician's clinical judgement
* able to communicate verbally in English and read English

Exclusion Criteria:

* unable to communicate verbally in English
* unable to read English
* cognitively unable to give informed consent (e.g. memory problems) as judged by referring physician or research assistant

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Advance care planning engagement | 12 weeks
  Survey measuring domains of engagement in advance care planning

SECONDARY OUTCOMES:
Advance care planning engagement-substitute decision maker | 12 weeks
  survey measuring substitute decision maker domains of engagement in advance care planning
Patient experience | 12 weeks
  survey of patient experience with intervention
Patient perceived impact on health care | 6-9 months
  qualitative interviews of patients asking perceived impact of intervention on later health care use

OTHER OUTCOMES:
Clinician experience of intervention | 6 months
  survey of clinician experience using conversation tools
Clinician confidence having advance care planning conversations | 6 months
  survey of clinician confidence, satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Howard, PhD, Principal Investigator — McMaster University
Locations (4):
- Canada (4):
  - Sunridge Family Medicine Teaching Centre, Calgary, Alberta
  - Safa Medical Clinic, Langley, British Columbia
  - New Westminster Family Practice, Vancouver, British Columbia
  - Vancouver General Hospital Gordon and Leslie Diamond Health Care Centre, Vancouver, British Columbia

REFERENCES:
- [Derived] Stevens J, Elston D, Tan A, Barwich D, Carter RZ, Cochrane D, Frenette N, Howard M. Clinicians' experiences implementing an advance care planning pathway in two Canadian provinces: a qualitative study. BMC Prim Care. 2024 Jun 15;25(1):217. doi: 10.1186/s12875-024-02468-4. PMID 38879532